CLINICAL TRIAL: NCT06635837
Title: Prospective Evaluation of the Role of Magnetic Resonance Imaging in Ovarian Masses During Pregnancy
Brief Title: Prospective Evaluation of the Role of MRI in Ovarian Masses During Pregnancy
Acronym: PROM-P
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6886
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian cancer represents 7% of all cancers in pregnant women. Characterizing an ovarian mass during pregnancy is essential to avoid unnecessary treatment and if treatment is required, to plan it accordingly. Ultrasound is the first line modality in these patients and various tools such as IOTA and ADNEX have been validated in non-pregnant patients to accurately categorize ovarian masses according to their malignant potential. A prospective multicentre study, in which Fondazione Policlinico Gemelli is involved, is currently ongoing aiming to validate these tools in pregnant Patients (p-IOTA).

Given the high contrast resolution and the absence of ionizing radiation, Magnetic Resonance Imaging is the preferred second-line modality. It increases the positive predictive value (PPV) of US from 7-50% to 70%, demonstrating a negative predictive value (NV) of 98%. In non-pregnant women, the Ovarian-Adnexal Reporting and Data System-MRI (ORADS-MRI) risk stratification system and the Non-Contrast MRI Score (NCMS) are commonly employed to assess the risk of malignancy in adnexal lesions with accuracies of 92% and 94%, respectively. Recently, both scoring systems have proven effective in retrospectively stratifying benign and malignant adnexal masses in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients > 18 years old
* Ability to understand and sign informed consent
* Patient with adnexal mass detected during pregnancy with either multilocular morphology or solid component at ultrasound examination
* Availability of MR imaging (1.5T and 3.0T MR scanner)
* Availability of histopathological reports obtained during pregnancy or within 3 months from delivery or at least one US follow-up examination 6-12 months after MRI examination

Exclusion Criteria:

* Patients lacking or with low quality MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with US-indeterminate adnexal masses detected during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the accuracy of MRI. | 5 years
  Evaluate the accuracy of MRI in discriminating benign versus malignant adnexal masses detected during pregnancy, by using subjective assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Panico, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Advanced Radiology Center- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No